CLINICAL TRIAL: NCT04212637
Title: Study of Eye Movements (EYE) as Early Markers of Brain Dysfunction (BRAIN) in Parkinson's Disease (PARK)
Acronym: eyebrainpark
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Laboratoire de Psychologie et NeuroCognition (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 38RC18.214
Record Dates: First submitted 2018-10-30; First posted 2019-12-27 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Volunteers (Experimental): MRI exam
  Interventions: Other: MRI
- Parkinson patient (Experimental): MRI exam
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — Examine BOLD activity in relation to eye movements measures
  Other Names: eyetracking

SUMMARY:
Identify the neural bases of eye movements during visual tasks and their dysfunction at early stages of Parkinson disease (de novo).

ELIGIBILITY:
Inclusion Criteria for all:

* Visual acuity normal or corrected to normal
* Affiliation to a social security scheme (copy of the vital card in support)
* Signed informed consent
* Medical examination according to the participation in the MRI examination
* MMSE score> 23/30

For Parkinson patient:

* Diagnosis of Parkinson's disease
* Presence of asymmetric bradykinesia and rest tremor and / or stiffness
* Hoehn & Yahr Stadium I-II / V

Exclusion Criteria for all:

* Unprotected Majors unable to express their consent
* Protected Major (Persons mentioned in Articles L1121-5,6 and 8 of the public health code)
* Significant hearing or motor impairment
* Past or present neuropsychiatric pathology (except benign epilepsy)
* Taking narcotics and / or drugs for neurocognitive purposes
* Existence of a severe condition in general (cardiac, respiratory, hematological, renal, hepatic, cancerous)
* Any other neurodegenerative pathology or treatment that may affect the oculomotor control

For Parkinson patient:

* Treatment for Parkinson's disease (except the inhibitors of monoaminoxidase B or MAO-B, such as selegiline and rasagiline).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
MRI images | 1 hour
  Functional and anatomical brain volumes

SECONDARY OUTCOMES:
Eye latency | 1 hour
  latency (milliseconds) of ocular saccades
eye amplitude | 1 hour
  amplitude (degree) of ocular saccades

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Grenoble-Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No